CLINICAL TRIAL: NCT02404025
Title: A Non-randomized, Phase II Study of Eltrombopag in Combination With Rabbit Anti-thymocyte Globulin/Cyclosporine A (ATG/CsA) in Subjects With Moderate or More Severe Aplastic Anemia Who Have Not Received Prior ATG/Anti-lymphocyte Globulin (ALG)-Based Immunosuppressive Therapy
Brief Title: Eltrombopag in Combination With Rabbit Anti-thymocyte Globulin/Cyclosporine A in Naive Aplastic Anemia (AA) Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 201793
Record Dates: First submitted 2015-02-26; First posted 2015-03-31 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Aplastic Anemia
Keywords: Eltrombopag; rabbit anti-thymocyte globulin; additive effect; cyclosporine A; bone marrow; hematopoietic stem cells; pancytopenia; leukopenia; platelets; throbocytopenia; mature blood cells; bone marrow biopsy
MeSH Terms: conditions — Anemia, Aplastic; Pancytopenia; Leukopenia | interventions — eltrombopag; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eltrombopag+rabbit ATG/CsA arm (Experimental): Subjects received rabbit ATG diluted by 500 mL of saline or 5% glucose injection at a dose of 2.5 to 3.75 mg per kilogram (kg) per day for 5 days as a slow intravenous infusion over 6 hours. CsA was administered at a dose of 3 mg per kg twice a day from day 0. The dose level was adjusted based on the monitoring of blood level or renal function. Eltrombopag was initiated on day 14 and it could be delayed up to 2 weeks if the subject had infection, serum sickness, or other adverse events. Eltrombopag wasadministered orally once a day at fasting at an initial dose of 75 mg, and the dose adjusted every 2 weeks according to the platelet count. Eltrombopag and CsA were continued until Week 26.After Week 26, eligible subjects received eltrombopag; and CsA was tapered or maintained as per the investigator's discretion.
  Interventions: Drug: Eltrombopag; Drug: Rabbit ATG; Drug: CsA

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag was provided as white round film-coated tablets containing 12.5 mg or 25 mg of eltrombopag free acid (SB-497115-GR, eltrombopag).
Drug: Rabbit ATG — Rabbit ATG, as an intravenous drip infusion, diluted by 500 mL of saline or 5% glucose injection was administered at a dose of 2.5 to 3.75 mg per kg per day as a slow intravenous infusion over 6 hours.
Drug: CsA — CsA as capsules, oral solution, or fine granule, was administered at a dose of 3 mg per kg twice a day.

SUMMARY:
This was an open label, non-randomized, phase II study of eltrombopag in combination with rabbit ATG/CsA in subjects with moderate or more severe AA who did not received prior ATG/ALG-based immunosuppressive therapy. The objective was to assess additive effects of eltorombopag on overall response rate (ORR) at 6 months (Week 26) of treatment with ATG/CsA. Subjects were assessed at least weekly for safety during the period from the start of ATG/CsA to 4 weeks after the start of administration of eltrombopag. After that, subjects had visits every 2 weeks until Week 26. Subjects in whom the treatment was assessed as effective at Week 26 could continued treatment with eltrombopag after 6 months when clinically indicated at the discretion of the investigator. There were five follow-up visits: at discontinuation of the treatment of eltrombopag, and Weeks 1, 2, 3, 4 and 26 after treatment discontinuation. As this study was the first Japanese phase II study in which this product was administered in combination with ATG/CsA to subjects with naive moderate or more severe AA, the subject number of this study was determined to be 10 based on the feasibility survey.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects aged >=18 and <71 years at the time of informed consent. Note: subjects aged >=71 and <75 may be eligible when clinically indicated at the discretion of the investigator by mutual agreement with Novartis medical advisor.
* Diagnosed with moderate or more severe AA according to the diagnostic criteria of AA. The severity classification is: Stage I - Mild - Other than the stages below; Stage II - Moderate - At least two of the following conditions are met: Reticulocyte <60,000/microliter, Neutrophil <1,000/microliter, Platelet <50,000/microliter; Stage III - Moderately severe - At least two of the following conditions are met and regular red blood cell transfusion (a need for transfusion of >=2 units per month) is required: Reticulocyte <60,000/microliter, Neutrophil <1,000/microliter, Platelet <50,000/microliter; Stage IV - Severe - At least two of the following conditions are met: Reticulocyte <20,000/microliter, Neutrophil <500/microliter, Platelet <20,000/microliter; Stage V - Very severe - At least one of the following conditions is met in addition to neutrophil <200/microliter: Reticulocyte <20,000/microliter, Platelet <20,000/microliter.
* Subjects who are considered an indication for the treatment with rabbit ATG and CsA.
* Adequate baseline organ function defined by the following criteria: Alanine aminotransferase (ALT), aspartate aminotransferase (AST)<=3 × local upper limit of normal (ULN) Creatinine, total bilirubin, and alkaline phosphatase (ALP) <1.5 × local ULN (total bilirubin <2.5 × local ULN with Gilbert's Syndrome)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0 or 1
* Subjects with QTcF<450 millisecond (msec) or QTcF<480 msec with branch block: QTc is QT interval corrected by Fridericia formula (QTcF), machine ,or manual overread. QTcF is based on single or averaged QTc value of triplicate ECG.
* Subjects are able to understand and comply with protocol requirements and instructions.
* Subjects have signed and dated informed consent.
* Subjects who meet one of the following conditions: Male subjects who have a female partner of childbearing potential must either have a prior vasectomy or agree to use an acceptable method of contraception from time of enrollment in the study until 16 weeks after the last dose of eltrombopag (based upon the lifecycle of sperm). Female subjects of non-childbearing potential (who are physiologically unable to become pregnant) defined as: Premenopausal women with documented bilateral oophorectomy, bilateral tubal ligation, or hysterectomy; or postmenopausal women after at least 12 months of natural amenorrhea [if uncertain, postmenopausal state should be confirmed by hematology result of follicle stimulating hormone (FSH) >40 milli-international units (mIU)/milliliter (mL) or estradiol <40 picogram (pg)/mL (<140 picomoles (pmol)/L)]. Female subjects of childbearing potential: Defined as those not meeting the definition of non-childbearing potential. Female subjects of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) or urine pregnancy test within 7 days prior to the first dose of ATG/CsA. It is recommended that the pregnancy test should be performed as close as possible to the first dose of ATG/CsA. Female subjects with a positive pregnancy test must be excluded from the study. Subjects with a negative pregnancy test must use acceptable contraception including abstinence after the pregnancy test. Subjects must agree to use the acceptable contraception including abstinence from 14 days prior to the first dose of ATG/CsA until 28 days after the last dose of eltrombopag.

Exclusion Criteria:

* Diagnosis of congenital AA (e.g. Fanconi anemia or Dyskeratosis congenital).
* Subjects who have a sibling donor with matched human leukocyte antigen (HLA) or who underwent hematopoietic stem cell transplantation (HSCT) previously. However, such subjects may be enrolled if HSCT is not indicated, or the subject does not want to undergo HSCT.
* Subjects with abnormal chromosome (monosomy 7 detected by fluorescence in situ hybridization (FISH), or other aberrations detected by G-band staining). Note: Subjects with abnormal chromosome which is not adopted into the clone definition of An International System for Human Cytogenetic Nomenclature (ISCN) may be enrolled after consulting with medical monitor.
* Previous ATG/ALG-based immunosuppressive therapy or steroid pulse therapy for AA.
* Treatment with CsA within 6 months before administration of ATG.
* Subjects with a paroxysmal nocturnal hemoglobinuria (PNH) clone size in granulocytes of >50% by flow cytometric analysis.
* Pre-existing cardiac disease (congestive heart failure New York Heart Association (NYHA) Grade II/III/IV), or arrhythmias known to involve the risk of thromboembolic events (e.g. atrial fibrillation)
* Past history of thromboembolic event (including anti-phospholipid antibody syndrome) and current use of anticoagulants.
* Subjects with past or current malignancy. Note : Subjects who have a history of completely resected malignant tumor and have been disease-free for 5 years are eligible.
* Subjects who test positive for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at screening.
* Infection not adequately responding to appropriate therapy.
* Subject with liver cirrhosis
* Subjects with any clinically significant severe cardiac, renal, or hepatic medical condition.
* Pregnant women (a positive serum or urine pregnancy test within 7 days prior to the first dose of ATG/CsA or lactating women) Note: Female subjects who are lactating are eligible to participate if they discontinue nursing prior to the first dose of ATG/CsA and refrain from nursing until 5 days after the completion of treatment with eltrombopag.
* Known hypersensitivity, intolerance or allergy to rabbit ATG, cyclosporine A, eltrombopag or any of their excipients.
* Current alcohol or drug abuse.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) proceeding the first dose of ATG/CsA.
* Subjects who is not candidates for ATG.
* Subjects who is not candidates for CsA.
* History of treatment with eltrombopag, romiplostim or other thrombopoietin-receptor (TPO-R) agonists.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Japan (8):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Ibaraki
  - Novartis Investigative Site, Ishikawa
  - Novartis Investigative Site, Miyagi
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Tochigi
  - Novartis Investigative Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subject started eltrombopag, and 1 subject was withdrawn from the study before starting eltrombopag, as he did not meet the eligibility criteria prior to receiving eltrombopag.
Groups:
- Eltrombopag+Rabbit ATG/CsA Arm: Subjects received rabbit ATG diluted by 500 mL of saline or 5% glucose injection at a dose of 2.5 to 3.75 mg per kilogram (kg) per day for 5 days as a slow intravenous infusion over 6 hours. CsA was administered at a dose of 3 mg per kg twice a day from day 0. The dose level was adjusted based on the monitoring of blood level or renal function. Eltrombopag was initiated on day 14 and it could be delayed up to 2 weeks if the subject had infection, serum sickness, or other adverse events. Eltrombopag was administered orally once a day at fasting at an initial dose of 75 mg, and the dose adjusted every 2 weeks according to the platelet count. Eltrombopag and CsA were continued until Week 26. After Week 26, eligible subjects received eltrombopag; and CsA was tapered or maintained as per the investigator's discretion.
Period: Overall Study
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Started | 10
Completed | 6
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] — Population: per protocol set
  years | 55.5 [39 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian Japanese | 10

OUTCOME MEASURES:

1. Primary Outcome: ORR at 6 Months: Overall Response Rate (ORR) Defined as the Number of Participants Who Met the Criteria of Either Complete Response (CR) or Partial Response (PR) at Week 26
Description: ORR will be calculated after 6 months of eltrombopag administration by measuring platelet, reticulocyte, neutrophil and transfusion independence. ORR includes Complete Response (CR) and Partial Response (PR) Rate.
Time Frame: Week 26
Population: Full analysis set; population obtained by excluding subjects: Eltrombopag was never administered to the subject during the study, subject had no baseline data: platelet count, hemoglobin, neutrophil count, and transfusion,subject had no data after the start of rabbit ATG therapy: platelet count, hemoglobin, neutrophil count, and transfusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Participants
  CR+PR | 7
  CR | 0
  PR | 7

2. Secondary Outcome: ORR at 3 Months
Description: ORR will be calculated after 3 months of eltrombopag administration by measuring platelet, reticulocyte, neutrophil and transfusion independence.
Time Frame: Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Participants | 2

3. Secondary Outcome: Complete Response (CR), and Partial Response (PR) Rate at 3 Months
Description: CR and PR will be calculated after 3 months of eltrombopag administration by measuring platelet, reticulocyte, neutrophil and transfusion independence.
Time Frame: Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Participants
  CR | 0
  PR | 2

4. Secondary Outcome: CR Rate Based on the Criteria Used in NIH 12-H-0150 Study at 6 Months
Description: CR criteria used in NIH 12-H-150 study is as follows: Hemoglobin >10 gram (g)/ deciliter (dL), and Absolute neutrophil count (ANC) >1,000/microliter, and Platelets >100,000/microliter.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Participants | 1

5. Secondary Outcome: Changes in Hematology Parameters (Haemoglobin) in the Absence of Platelet Transfusion
Description: The change in hematology values ( haemoglobin) were evaluated.
Time Frame: Week 26 and week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
g/L
  Haemoglobin changes from baseline, week 26 (g/L): number analyzed (Participants) | 9
  Haemoglobin changes from baseline, week 26 (g/L) | 24.6 (19.20)
  Haemoglobin changes from baseline, week 104 (g/L): number analyzed (Participants) | 3
  Haemoglobin changes from baseline, week 104 (g/L) | 39.0 (3.61)

6. Secondary Outcome: Changes in Hematology Parameters in the Absence of Platelet Transfusion
Description: The change in hematology values from baseline for platelets, neutrophils and reticulocytes were evaluated.
Time Frame: Week 26 and week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gi/L
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Gi/L
  neutrophils changes from baseline, week 26 (Gi/L): number analyzed (Participants) | 9
  neutrophils changes from baseline, week 26 (Gi/L) | 1.2196 (0.59501)
  neutrophils changes from baseline, week 104 (Gi/L): number analyzed (Participants) | 3
  neutrophils changes from baseline, week 104 (Gi/L) | 1.2978 (0.65819)
  platelets changes from baseline, week 26 (Gi/L): number analyzed (Participants) | 9
  platelets changes from baseline, week 26 (Gi/L) | 66.94 (57.187)
  platelets changes from baseline, week 104 (Gi/L): number analyzed (Participants) | 3
  platelets changes from baseline, week 104 (Gi/L) | 107.33 (4.041)
  reticulocytes changes from baseline week 26 (Gi/L): number analyzed (Participants) | 8
  reticulocytes changes from baseline week 26 (Gi/L) | 30.0175 (21.81519)
  reticulocytes changes from baseline week104 (Gi/L): number analyzed (Participants) | 2
  reticulocytes changes from baseline week104 (Gi/L) | 48.0900 (29.96719)

7. Secondary Outcome: Frequency of Platelet and Red Blood Cells (RBC) Transfusions
Description: RBC transfusion dependency defined as at least one RBC transfusion within 8 weeks prior to D1. Platelet or RBC transfusions will be based on physician's subjective judgement. Platelet transfusion will be done if the platelet count is less than 10×10^9/liter (L) with significant bleeding tendency or the platelet count is less than 20×10^9/L with pyrexia. RBC transfusion will be done to keep the hemoglobin concentration at over 7 g/dL or in the presence of clinical symptoms such as dyspnea.
Time Frame: Baseline, Week 26
Population: full analysis set, participants who were transfusion dependant
Measure: Mean (Standard Deviation); unit: mean of transfusions number
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
mean of transfusions number
  Baseline RBC transfusions | 4.0 (3.10)
  Week 26 RBC transfusions: number analyzed (Participants) | 5
  Week 26 RBC transfusions | 1.0 (2.24)
  Baseline Platelet transfusion: number analyzed (Participants) | 8
  Baseline Platelet transfusion | 3.4 (2.77)
  Week 26 Platelet transfusion: number analyzed (Participants) | 7
  Week 26 Platelet transfusion | 1.0 (1.91)

8. Secondary Outcome: Volume of Platelet and RBC Transfusions
Description: Platelet or RBC transfusions will be based on physician's subjective judgement. Platelet transfusion will be done if the platelet count is less than 10×10^9/L with significant bleeding tendency or the platelet count is less than 20×10^9/L with pyrexia. RBC transfusion will be done to keep the hemoglobin concentration at over 7 g/dL or in the presence of clinical symptoms such as dyspnea.
Time Frame: Baseline, Week 26
Population: Full analysis set, patients who were transfusion dependent
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
mL
  Baseline RBC transfusion | 1600.0 (1239.35)
  Week 26 RBC transfusion | 400.0 (894.43)
  Baseline Platelet transfusion: number analyzed (Participants) | 8
  Baseline Platelet transfusion | 687.5 (559.18)
  Week 26 Platelet transfusion: number analyzed (Participants) | 7
  Week 26 Platelet transfusion | 200.0 (382.97)

9. Secondary Outcome: The Proportion of Subjects Whose Transfusion Unit (or Volume) Are Decreased or Who Became Transfusion (Platelet, RBC) Independent
Description: The proportions of the subjects for whom the amount of blood transfusion (platelets and RBC) decreased or the proportions of the subjects for whom blood transfusion (platelets and RBC) became unnecessary. Platelet transfusion will be done if the platelet count is less than 10×10^9/L with significant bleeding tendency or the platelet count is less than 20×10^9/L with pyrexia. RBC transfusion will be done to keep the hemoglobin concentration at over 7 g/dL or in the presence of clinical symptoms such as dyspnea.
Time Frame: Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Participants
  Baseline RBC transfusion dependence | 6
  RBC Transfusion decrease or free | 4
  Baseline Platelet transfusion dependence | 8
  Platelet Transfusion decrease or free | 5

10. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization is the time period from the administration of ATG up to discharge.
Time Frame: Week 26
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
days | 49.0 [13 to 123]

11. Secondary Outcome: Time to Onset of CR and PR
Description: The time to onset of CR and PR will be determined by measuring platelet, reticulocyte, neutrophil and transfusion independence.
Time Frame: Week 26
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
months | 3.75 [2.5 to 4.8]

12. Secondary Outcome: Duration of CR or PR
Description: Duration for CR or PR will be determined by measuring platelet, reticulocyte, neutrophil and transfusion independence.
Time Frame: Week 104
Population: Number of participants who responded to treatment (7 out of the 10 participants)
Measure: Median (Full Range); unit: months
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 7
months | 17.28 [6.0 to 20.3]

13. Secondary Outcome: Degree of Exposure to Eltrombopag : Average Daily Dose
Time Frame: Week 104
Population: safety population:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
mg/day | 43.8 (23.19)

14. Secondary Outcome: Degree of Exposure to Eltrombopag : Cumulative Dose
Description: The cumulative dose of drug administered to the subject will be calculated.
Time Frame: Week 104
Population: safety population:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
mg | 17687.5 (7179.77)

15. Secondary Outcome: Degree of Exposure to Eltrombopag : Days on Study
Time Frame: Week 104
Population: safety population:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
days | 493.7 (233.69)

16. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be collected from the start of study treatment until the approval.
Time Frame: though study completion , approximately 2 years
Population: safety population:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Participants
  number of participants with an AE | 10
  with an AE related to any study treatment | 8
  with an AE related to Eltrombopag | 5
  with an AE related to CsA | 8
  number of participants with a SAE | 2

17. Secondary Outcome: Vital Signs (Blood Pressure) as a Measure of Safety and Tolerability
Description: Vital sign measurements : blood pressure
Time Frame: baseline and Week 26
Population: safety set:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
mmHg
  baseline systolic blood pressure (mmHg) | 115.7 (15.06)
  week 26 systolic blood pressure (mmHg): number analyzed (Participants) | 9
  week 26 systolic blood pressure (mmHg) | 126.4 (17.12)
  baseline diastolic blood pressure (mmHg) | 64.3 (11.78)
  week 26 diastolic blood pressure (mmHg): number analyzed (Participants) | 9
  week 26 diastolic blood pressure (mmHg) | 76.9 (13.11)

18. Secondary Outcome: 12-lead Electrocardiogram (ECG) as Measure of Safety and Tolerability
Description: Triplicate 12-lead ECGs will be obtained at designated time points during the study using an ECG machine that calculates the heart rate and measures PR, QRS, QT, and QT interval corrected by Fridericia formula (QTcF) intervals.
Time Frame: Baseline, Week 26
Population: safety population: The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Participants
  screening (baseline): normal | 8
  screening (baseline): abnormal not clinically significant | 2
  screening (baseline): abnormal clinically significant | 0
  week 26: number analyzed (Participants) | 9
  week 26: normal | 6
  week 26: abnormal not clinically significant | 3
  week 26: abnormal clinically significant | 0

19. Secondary Outcome: The Trough Concentrations of Eltrombopag Following Repeat Doses of at 75 mg, 50 mg and 25 mg
Description: Blood samples will be collected after repeat (14 days) doses of eltrombopag 75, 50, 25 mg to determine the plasma eltrombopag concentration prior to the next dose.
Time Frame: day 15
Population: pharmacokinetic population:The PK population was defined as all subjects whose PK samples were collected and measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
ng/mL
  Eltrombopag 25 mg day 15, 0h (predose): number analyzed (Participants) | 1
  Eltrombopag 25 mg day 15, 0h (predose) | 6070 (NA) — only 1 measure (from 1 participant) at that dose level
  Eltrombopag 50 mg day 15, 0h (predose): number analyzed (Participants) | 2
  Eltrombopag 50 mg day 15, 0h (predose) | 20800 (7920)
  Eltrombopag 75 mg day 15, 0h (predose) | 21800 (7370)

20. Secondary Outcome: The Concentration After 4 Hours of Dose of Eltrombopag 75 mg
Description: Blood sample will be collected at 4 hours after repeat (14 days) dose of eltrombopag 75 mg
Time Frame: day 15
Population: pharmacokinetic population: The PK population was defined as all subjects whose PK samples were collected and measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
ng/mL
  day 15, 0 hour (predose) | 21800 (7370)
  day 15, 4 hours (post dose) | 28400 (8960)

21. Secondary Outcome: Composite of Laboratory Parameters Assessment as a Safety Measure (Haemoglobin and Albumin).
Description: The laboratory test values (haemoglobin and albumin) were calculated at each time point of evaluation.
Time Frame: Baseline, Week 26
Population: safety set:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
g/L
  hemoglobin baseline (g/L) | 77.2 (4.52)
  hemoglobin week 26 (g/L): number analyzed (Participants) | 9
  hemoglobin week 26 (g/L) | 102.4 (17.64)
  Albumin baseline (g/L) | 38.7 (4.83)
  Albumin Week 26 (g/L): number analyzed (Participants) | 9
  Albumin Week 26 (g/L) | 44.9 (2.52)

22. Secondary Outcome: Composite of Laboratory Parameters Assessment as a Safety Measure (Lymphocytes and Neutrophils).
Description: The laboratory test values (lymphocytes and neutrophils) were calculated at each time point of evaluation.
Time Frame: Baseline, Week 26
Population: safety set:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: Gi/L
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
Gi/L
  White blood cell count baseline (Gi/L) | 1.896 (0.9200)
  White blood cell count week 26(Gi/L): number analyzed (Participants) | 9
  White blood cell count week 26(Gi/L) | 2.682 (0.8347)
  lymphocytes baseline (Gi/L) | 1.3943 (0.60771)
  lymphocytes week 26 (Gi/L): number analyzed (Participants) | 9
  lymphocytes week 26 (Gi/L) | 0.7108 (0.34079)
  Total Neutrophils Baseline (Gi/L) | 0.4033 (0.38230)
  Total Neutrophils Week 26 (Gi/L): number analyzed (Participants) | 9
  Total Neutrophils Week 26 (Gi/L) | 1.6120 (0.468)

23. Secondary Outcome: Composite of Laboratory Parameters Assessment as a Safety Measure (Alcaline Phosphatase and Aspartate Amino Transferase) .
Description: The laboratory test values (Alcaline Phosphatase and Aspartate Amino Transferase) were calculated at each time point of evaluation.
Time Frame: Baseline, Week 26
Population: safety set:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
IU/L
  Alcaline phosphatase baseline (IU/L) | 186.7 (57.03)
  Alcaline phosphatase Week 26 (IU/L): number analyzed (Participants) | 9
  Alcaline phosphatase Week 26 (IU/L) | 319.6 (114.58)
  Alanine Amino Transferase baseline (IU/L) | 14.3 (3.71)
  Alanine Amino Transferase Week 26(IU/L): number analyzed (Participants) | 9
  Alanine Amino Transferase Week 26(IU/L) | 16.8 (7.48)
  Aspartate Amino Transferase baseline (IU/L) | 14.9 (2.47)
  Aspartate Amino Transferase Week 26(IU/L): number analyzed (Participants) | 9
  Aspartate Amino Transferase Week 26(IU/L) | 18.8 (4.66)

24. Secondary Outcome: Composite of Laboratory Parameters Assessment as a Safety Measure.
Description: The laboratory test values (hematological /biochemical examinations) were calculated at each time point of evaluation.
Time Frame: Baseline, Week 26
Population: safety set:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
umol/L
  Direct Bilirubin baseline (umol/L) | 2.565 (0.9012)
  Direct Bilirubin week 26 (umol/L): number analyzed (Participants) | 9
  Direct Bilirubin week 26 (umol/L) | 2.850 (1.2092)
  Indirect Bilirubin baseline (umol/L) | 5.301 (2.2002)
  Indirect Bilirubin week 26 (umol/L): number analyzed (Participants) | 9
  Indirect Bilirubin week 26 (umol/L) | 6.080 (1.7336)
  Total Bilirubin baseline (umol/L) | 7.866 (2.9287)
  Total Bilirubin week 26 (umol/L): number analyzed (Participants) | 9
  Total Bilirubin week 26 (umol/L) | 8.930 (2.5331)
  Creatinine baseline (umol/L) | 59.6700 (11.86193)
  Creatinine week 26 (umol/L): number analyzed (Participants) | 9
  Creatinine week 26 (umol/L) | 79.9529 (23.55122)
  Potassium baseline (umol/L) | 3.88 (0.371)
  Potassium week 26 (umol/L): number analyzed (Participants) | 9
  Potassium week 26 (umol/L) | 4.27 (0.335)
  Sodium baseline (umol/L) | 140.7 (1.42)
  Sodium week 26 (umol/L): number analyzed (Participants) | 9
  Sodium week 26 (umol/L) | 140.4 (1.74)

25. Secondary Outcome: Vital Signs (Temperature) as a Measure of Safety and Tolerability
Description: Vital sign measurements : temperature
Time Frame: baseline and Week 26
Population: safety set:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
°C
  baseline temperature (°C) | 36.55 (0.448)
  week 26 temperature (°C): number analyzed (Participants) | 9
  week 26 temperature (°C) | 36.71 (0.379)

26. Secondary Outcome: Vital Signs (Pulse Rate) as a Measure of Safety and Tolerability
Description: Vital sign measurements : pulse rate.
Time Frame: baseline and Week 26
Population: safety set:The safety population consisted of all subjects who received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Eltrombopag+Rabbit ATG/CsA Arm
Number analyzed (Participants) | 10
beats/min
  baseline heart rate (beats /min) | 76.2 (10.38)
  week 26 heart rate (beats/min): number analyzed (Participants) | 9
  week 26 heart rate (beats/min) | 80.4 (10.82)

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse events are reported in this record from First Patient First Treatment until Last Patient Last Visit up to approximately 2 years.
Description: AE additional description
Groups:
- Eltrombopag+ATG/CsA: Eltrombopag+ATG/CsA
Arm/Group | Eltrombopag+ATG/CsA
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag+ATG/CsA (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag+ATG/CsA (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Dry eye (Eye disorders) | 2
Chronic gastritis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Epstein-Barr virus infection (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 1
Oral infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Amylase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 1
Cytomegalovirus test positive (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Serum ferritin increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Iron overload (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Paralysis (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis'agreements with its investigators may vary. However Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.